CLINICAL TRIAL: NCT01925677
Title: Use of the Intuitive Surgical da Vinci® Single-Site™ With Instruments and Accessories for Single-Port Laparoscopic Nephrectomies
Brief Title: Robotic Single Port Donor Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Rolf Barth, Director of Liver Transplantation, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00055955
Record Dates: First submitted 2013-08-06; First posted 2013-08-20 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Renal Transplant Donor of Left Kidney; Donor Nephrectomy; Robotic Surgery; Single-port
Keywords: Transplant; donor; nephrectomy; robotic; laparoscopy; single-port

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- da Vinci® Single-Site™ (Experimental): Robotic-assisted single-incision laparoscopic nephrectomy.
  Interventions: Device: da Vinci® Single-Site™

INTERVENTIONS:
Device: da Vinci® Single-Site™ — Planned single-incision laparoscopic nephrectomy performed with the assistance of the Da Vinci Robotic Surgical System.

SUMMARY:
Feasibility study on robotic-assisted single-site donor nephrectomy utilizing da Vinci instrumentation and Single-Site platforms.

DETAILED DESCRIPTION:
Our center has performed over 200 single-port donor nephrectomies with standard laparoscopy and has reported patient benefits associated with a single port approach. The single port robotic platform offers the potential to ameliorate the significant technical and ergonomic challenges that currently limit more widespread application of single port donor surgery. After being informed of the potential risks and off-label use of the da Vinci Single-Site approach in our study, patients will undergo a robotic-assisted single-site donor nephrectomy performed by a two-surgeon team utilizing existing da Vinci instrumentation and Single-Site platforms. Renal mobilization and vascular dissection will be performed with manual laparoscopy performed for vascular division utilizing stapling devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be approved by the Living Donor Center.
* Patient must have compatible blood type with the recipient.
* Patient must have body mass index less than 35.
* Patient must have appropriate anatomy for left kidney donation.

Exclusion Criteria:

* Any patient receiving anticoagulant drugs such as Coumadin or warfin
* Any patient suffering from an active urinary tract infections
* Any patients suffering from cancer.
* Any patients suffering from diabetes.
* Any patients suffering from kidney disease.
* Any patients suffering from heart disease.
* Any patients suffering from liver disease.
* Any patients suffering from HIV or hepatitis
* Any patients suffering from previous major abdominal surgery.
* Any patients suffering from more than two left renal arteries.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf N Barth, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barth RN, Phelan MW, Goldschen L, Munivenkatappa RB, Jacobs SC, Bartlett ST, Philosophe B. Single-port donor nephrectomy provides improved patient satisfaction and equivalent outcomes. Ann Surg. 2013 Mar;257(3):527-33. doi: 10.1097/SLA.0b013e318262ddd6. PMID 22968070

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | da Vinci® Single-Site™
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | da Vinci® Single-Site™
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 52 [42 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Caucasian | 3
Region of Enrollment [Number; unit: participants]
  United States | 3
Number of participants [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Successful Completion of the Surgical Procedure
Description: The primary objective is to determine the feasibility measure of the current Single-Site platform to perform donor nephrectomy prior to vascular division and extraction. Specifically, it will be recorded which portions of the operation utilized the robotic device. The primary outcome variable is the completion of the operation for kidney donation.
Time Frame: during operation
Measure: Count of Participants; unit: Participants
Arm/Group | da Vinci® Single-Site™
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Operative Times
Description: Operative times will closely be measured
Time Frame: during operation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | da Vinci® Single-Site™
Number analyzed (Participants) | 3
minutes | 82 (16)

3. Secondary Outcome: Blood Loss
Description: Blood loss of patients will be closely monitored and recorded.
Time Frame: during operation
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | da Vinci® Single-Site™
Number analyzed (Participants) | 3
mL | 77 (64)

4. Secondary Outcome: The Comparison of Surgeon Ergonomic Questionnaires in Robotic Assisted Versus Standard Laparoscopic Single Port Donor Nephrectomies.
Description: A surgeon ergonomics questionnaire will be given to surgeons after performing both robotic assisted and standard laparoscopic single port donor nephrectomies. The results from both of these surveys will then be compared. These are qualitative and were not analyzed for statistical trends.
Time Frame: intra-operative experience collected within 24 hours
Population: surgeon questionnaire
Measure: Number; unit: participants
Arm/Group | da Vinci® Single-Site™
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Time Frame: Data was collected for 1 year from time of surgery
Arm/Group | da Vinci® Single-Site™
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT01925677/Prot_SAP_000.pdf